CLINICAL TRIAL: NCT01325454
Title: Angiogenic Cytokines and Fibrinolytic Activity in Parapneumonic Effusions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chi-Li Chung MD, PhD, Division of Pulmonary Medicine, Department of Internal Medicine,Taipei Medical University Hospital
Other Study IDs: TMUH-PARAPNEUMONIC STUDY
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Pleural Effusion
Keywords: Pleural effusion; angiogenic cytokine; fibrinolytic activity
MeSH Terms: conditions — Pleural Effusion | interventions — Chest Tubes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pleural effusions
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with parapneumonic effusions: Patients with pleural effusions of unknown causes admitted to Taipei Medical University Hospital were included if parapneumonic effusion was diagnosed as one associated with pneumonia according to the criteria of the American Thoracic Society (ie, patients with newly acquired respiratory symptoms, fever, and abnormal breath sounds, plus a new lung infiltrate seen on a chest radiograph).
  Interventions: Device: pleural pigtail drainage

INTERVENTIONS:
Device: pleural pigtail drainage — With the guidance of chest US, 50 ml of pleural fluid was collected using a standard thoracentesis technique immediately or within 24 hr after hospitalization. When pleural effusion was multi-loculated, the fluid was aspirated from the largest loculus. Routine analyses of pleural fluid for total leukocytes, cell differentials of leukocytes, pH value, and levels of protein, glucose and LDH were performed in addition to cytological and microbiologic examination of pleural fluid.The rest of pleural fluid samples were mixed with 3.8 % sodium citrate in a 9:1 ratio of pleural fluid to citrate. The sodium citrate-mixed pleural fluid specimens were immersed in ice immediately and then centrifuged at 2,500 g for 10 minutes. The cell-free supernatants of pleural fluid were frozen at -70℃ immediately after centrifuge for later measurements. The commercially available enzyme-linked immunosorbent assay kits were used to measure the effusion levels of VEGF, IL-8 , tPA and PAI-1.
  Other Names: chest drain; chest tube drainage; tube thoracostomy

SUMMARY:
Angiogenesis is a key process in the formation of exudative pleural effusions. Fluid loculation is common in parapneumonic effusion and is associated with depressed pleural fibrinolytic activity and poor clinical outcome. However, the relationship between angiogenic cytokines and fibrinolytic activity in the pleural space remains unclear. The researchers's hypothesis is that the levels of angiogenic cytokines were increased and associated with decreased fibrinolytic activity in parapneumonic effusions which may contribute to fibrin deposition and fluid loculation in the pleural space.

DETAILED DESCRIPTION:
Formation of parapneumonic effusions (PPE) involves increased pleural vascular permeability induced by the contiguous pneumonia. It has been demonstrated that exposure of pleural mesothelial cells to bacteria or lipopolysaccharide (LPS) leads to increased release of angiogenic factors, including vascular endothelial growth factor (VEGF) and interleukin (IL)-8, which induce vascular hyperpermeability, fluid exudation, and neutrophil influx into the pleural space, and may play a pivotal role in development of PPE. With persistent inflammation and angiogenesis, amplified vascular and mesothelial permeability leads to increased plasma extravasation, activation of the coagulation cascade, and repression of fibrinolytic activity within the pleural cavity, which contribute to the development of a ''complicated'' PPE, manifested with fibrin deposition and pleural fluid loculation. Fibrin turnover in the pleural cavity is greatly affected by fibrinolytic activity mediated by plasmin, which is regulated mainly by the equilibrium between plasminogen activators (PAs) and plasminogen activator inhibitors (PAIs).VEGF induces vascular hyperpermeability and may facilitate the genesis of fibrin gel in PPE. Previous studies reported that VEGF plays a role in the modulation of tPA and PAI-1, and that anti-VEGF antibody attenuates pleurodesis induced by transforming growth factor-β2. These findings suggest that VEGF may be involved in the regulation of fibrin turnover, fluid loculation and tissue fibrosis in the pleural space. Enhanced procoagulant and depressed fibrinolytic activities have been observed in PPE. However, the relationship between angiogenic cytokines and fibrinolytic activity in PPE remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pleural effusions of unknown causes admitted to Taipei Medical University Hospital were included if parapneumonic effusion was diagnosed as one associated with pneumonia according to the criteria of the American Thoracic Society (ie, patients with newly acquired respiratory symptoms, fever, and abnormal breath sounds, plus a new lung infiltrate seen on a chest radiograph).

Exclusion Criteria:

* History of chest trauma or invasive procedures directed into the pleural cavity; bleeding disorder or anticoagulant therapy
* Use of streptokinase in the previous 2 years; and likely survival less than 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pleural effusions of unknown causes admitted to Taipei Medical University Hospital were included.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Response to treatment including improvement in vital signs and chest radiography | 5 days after treatment within admission

SECONDARY OUTCOMES:
Chest radiography and pulmonary function testing with spirometry. | At discharge, and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Li Chung, MD, PhD, Principal Investigator — Division of Pulmonary Medicine, Taipei Medical University, Taipei, Taiwan
Locations (1):
- Division of Pulmonary Medicine, Taipei Medical University Hospital, Taipei, Taiwan